CLINICAL TRIAL: NCT06758765
Title: Comparison of the Effects of the Erector Spinae Plane Block and PECS I-II Blocks on Postoperative Opioid Consumption and Pain Scores of Patients After Breast-conserving Surgery: A Prospective Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block vs. PECS I-II Blocks After Breast-conserving Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Taner Abdullah, Principal Investigator, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022.02.44
Record Dates: First submitted 2024-12-20; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Surgery; Breast Conserving Surgery; Erector Spinae Plane Block; Pectoral Nerve (PECS) Block; Visual Analog Scale; Opioid Consumption; Postoperative Pain, Acute
Keywords: erector spinae plane block; pectoral nerve (PECS) block; postoperative pain; breast conserving surgery
MeSH Terms: conditions — Bites and Stings; Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP group (Experimental): The group that received erector spinae plane block
  Interventions: Procedure: Erector Spinae Plane Block
- PECS group (Experimental): The group that received PECSI-II blocks
  Interventions: Procedure: Pectoral Nerve Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — ESPB was applied to the patients in a sitting position. A high-frequency linear probe was used. Under sterile conditions, the USG probe was placed longitudinally approximately 2 cm lateral to the T4 spinous process. Skin, subcutaneous fat tissue, m. trapezius, rhomboid muscles, erector group muscles, transverse process, intercostal muscles, pleura and lung movements were visualized from superficial to deep structures. 1 ml of 2% lidocaine was injected into the estimated needle entry area. Then, with the block needle the m. trapezius, mm. rhomboidei and erector spinae muscles were passed in order with the in-plane method and the needle was brought into contact with the transverse process. Fascial separation was confirmed with 1-2 ml of saline solution and the block was performed by injecting 20 ml of 0.375% bupivacaine. The distribution of the drug was confirmed by observing it with USG.
  Arms: ESP group
Procedure: Pectoral Nerve Block — The PECSI and PECSII blocks were applied concurrently.
  In patients who will undergo PECS II, sterile conditions were prepared with the arm on the side to be operated on in the supine position and 90 degrees of abduction. The lateral and pectoral branches of the thoracoacromial artery were visualized between the PM and Pm muscles at the level of the 4th rib under USG guidance. The blocking needle was directed between the PM and Pm muscles for PECS I, 1-2 ml of saline was injected to verify fascial spread, and 10 ml of 0.375% bupivacaine was applied. Afterwards, fascial spread was confirmed by injecting 1-2 ml of saline between the pectoralis minor muscle and the serratur anterior muscle, and PECS II was performed by injecting 10 ml of 0.375% concentration bupivacaine. The distribution of the drug was confirmed by observing it with USG.
  Arms: PECS group

SUMMARY:
The goal of this study is to compare the analgesic effects of ESPB and PECS II blocks in patients undergoing BCS. The main question it aims to answer is:

* Whether these two different block procedures will create a difference in postoperative pain scores.
* Comparison of total opioid consumption during the 24-hour postoperative period.

Our study included patients who were female, who were going to undergo elective breast-conserving surgery between March 2022 and August 2022.

DETAILED DESCRIPTION:
The patients to be included in our study were divided into two groups as ESPB group or PECS II group by an anesthesia assistant independent of the study using a computer-based randomization program one day before the operation. All patients were informed about the block in the preoperative period, the use of the patient-controlled analgesia device to be used after the operation, and Visual Analog Scale (VAS) assessment. (Patients were asked to indicate their pain on a scale where 0 represented "no pain" and 10 represented "unbearable pain.)

On the day of the operation, group envelopes were placed in the patient files to indicate the groups in sealed envelopes. The appropriate anesthesia method was applied to the patient according to the group written on the patient's envelope by the relevant anesthesiologist on duty in the study. Our study was conducted as a randomized controlled and prospective study.

VAS scores at 0, 15, 30, 60 minutes postoperatively recorded for the primer output of the study. For the secondary outputs the total amount of analgesic used was recorded from the records of the PCA device. All patients' demographic data, intraoperative hemodynamic data, anesthesia duration, surgical duration and hospital stay, VAS at 4, 6, 12, 24 hours in the service follow-up, rescue analgesic requirements and numbers, nausea-vomiting and developing complications were evaluated and recorded. The evaluations were made by the anesthesiologist who was blind to the groups.

ELIGIBILITY:
Inclusion Criteria:

* female
* age between 18-70
* underwent breast conserving surgery

Exclusion Criteria:

* patients with coagulopathy
* known local anesthetic allergy
* abnormal liver function tests
* infection at the planned injection site
* chronic usage of analgesics
* under the age of 18
* over the age of 70
* ASA (American Society of Anesthesiologists) IV and higher risk classes
* limited cooperation for Visual Analog Scale (VAS) follow-ups

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because breast cancer is very rare in men
Enrollment: 72 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Early postoperative Visual Analog Scale (VAS) scores | First hour after surgery
  The postoperative pain level that evaluated with evaluated with VAS at 0, 15, 30 and 60 minutes.
  Patients were asked to indicate their pain on a scale where 0 represented "no pain" and 10 represented "unbearable pain".

SECONDARY OUTCOMES:
Additional opioid analgesic requirement in the postanesthesia care unit | First hour after surgery
  Patients who scored 4 and above in the pain score were administered 10 mg meperidine.
Total opioid consumption after discharging from postanesthesia care unit | Between 1-24 hours after surgery
  The PCA device, which was applied to the patients at the 60th minute postoperatively, was left for patient use until the 24th hour postoperatively.
Visual Analog Scale (VAS) during 24 hours follow-up after surgery | 1th, 4th, 6th, 12th, and 24th hours postoperatively
  VAS values after discharge from the postanesthesia care unit
  Patients were asked to indicate their pain on a scale where 0 represented "no pain" and 10 represented "unbearable pain".

CONTACTS AND LOCATIONS:
Overall Officials: Funda Gümüş Özcan, Prof, Study Chair — Basaksehir Cam ve Sakura State Hospital
Locations (1):
- Basaksehir Cam ve Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bakeer A, Abdallah NM. Erector Spinae Plane Block Versus PECS Block Type II for Breast Surgery: A Randomized Controlled Trial. Anesth Pain Med. 2022 Apr 25;12(2):e122917. doi: 10.5812/aapm-122917. eCollection 2022 Apr. PMID 35991781
- [Result] Hong B, Bang S, Oh C, Park E, Park S. Comparison of PECS II and erector spinae plane block for postoperative analgesia following modified radical mastectomy: Bayesian network meta-analysis using a control group. J Anesth. 2021 Oct;35(5):723-733. doi: 10.1007/s00540-021-02923-x. Epub 2021 Mar 30. PMID 33786681
- [Result] Altiparmak B, Korkmaz Toker M, Uysal AI, Turan M, Gumus Demirbilek S. Comparison of the effects of modified pectoral nerve block and erector spinae plane block on postoperative opioid consumption and pain scores of patients after radical mastectomy surgery: A prospective, randomized, controlled trial. J Clin Anesth. 2019 May;54:61-65. doi: 10.1016/j.jclinane.2018.10.040. Epub 2018 Nov 3. PMID 30396100